CLINICAL TRIAL: NCT07391189
Title: Study on the Health Effects of Adapted Physical Activity From Japanese Martial Arts-Aikido.
Brief Title: Healthy Effects of Adapted Aikido in People With Grip Disfunction
Acronym: AdAikido
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Francisco Javier López Román, Investigator, Universidad Católica San Antonio de Murcia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCAMCFE-00042
Record Dates: First submitted 2026-01-29; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Unilateral Handgrip Dysfunction
Keywords: Aikido; Handgrip Dysfunction; Adapted Physical Activity; Exercise Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Case group (Experimental): Case group is formed by people with handgrip dysfunction
  Interventions: Other: Participation in an adapted aikido program
- Control group (Active Comparator): Control group is formed by healthy people
  Interventions: Other: Participation in an adapted aikido program

INTERVENTIONS:
Other: Participation in an adapted aikido program — The aikido program has been adapted for optimal practice by people with handgrip dysfunction. Several key components of the techniques have been modified to enable their performance by individuals with limited hand mo- bility.

SUMMARY:
This study investigates the effects of an adapted aikido exercise program on

the health of adults with unilateral wrist and/or hand dysfunction. The un- derlying assumption is that regular practice of adapted aikido may improve

physical, psychological, and quality-of-life parameters in this population com- pared with a non-exercising control group.

DETAILED DESCRIPTION:
The primary objective is to assess the physical health benefits derived from an adapted aikido training program in people with unilateral reduction of wrist and hand functionality. Secondary objectives are to examine poten- tial benefits on mental health and to evaluate the influence of aikido practice on quality of life. Accordingly, the working hypothesis is that participation in the program will lead to significant improvements in physical, functional, and psychological variables compared with the control group.

A longitudinal, controlled, single-center study with repeated measures is proposed, including 20 adult participants, 10 in the intervention group and 10 in the control group, all without prior aikido experience and not practicing other martial arts during the study. The intervention consists of an adapted aikido program with two one-hour sessions per week over approximately four months, delivered by an experienced instructor, with systematic attendance recording to monitor adherence.

Primary outcomes include arm muscle mass, muscle strength (analytical dynamometry and handgrip test), active range of motion of the wrist, el- bow, and shoulder, body mass index, and cardiac function assessed via heart rate during exercise. Secondary outcomes are upper limb function (DASH), pain (VAS), sleep quality (PSQI and accelerometry), body awareness (BAQ), mindfulness (MAAS), anxiety (Hamilton Anxiety Scale), and positive and negative affect (PANAS).

Assessments will be conducted at three time points (baseline, mid-intervention, and post-intervention), combining clinical history, physical measurements, heart rate recordings, and psychological and quality-of-life questionnaires. Statistical analysis will include descriptive statistics, tests for normality and homoscedasticity, and repeated-measures ANCOVA with a significance level of 0.05 using R software, to determine the effect of adapted aikido on the different health indicators.

ELIGIBILITY:
Inclusion Criteria:

* Be of legal age.
* Have no prior knowledge of aikido.
* Not be practicing other martial arts at the time of inclusion in the study or during the adapted training program.
* Unilateral dysfunction of the hand and/or wrist that prevents or hinders tasks related to gripping (only for case group).

Exclusion Criteria:

* Presence of anatomical or functional alterations that could affect the performance of aikido techniques (other than those allowed for the study group).
* Intellectual disability and/or inability to understand the informed con- sent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01-19 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-07-15 (Estimated)

PRIMARY OUTCOMES:
Arm muscle mass | The evolution of the variable will be evaluated on days 60 and 120.
  Estimated from arm circumference and triceps skinfold measurements. The instruments used will be an anthropometric tape and a skinfold caliper, respectively.
Muscle strength | The evolution of the variable will be evaluated on days 60 and 120.
  Analytical strength measurements will be taken for the main muscles responsible for each movement of the upper limb, as well as a handgrip test to assess overall hand grip strength. The instruments used will be a Jamar dynamometer and a hand-held dynamometer.
Active joint mobility of the wrist, elbow, and shoulder | The evolution of the variable will be evaluated on days 60 and 120.
  It will be measured using a digital inclinometer, an instrument that has shown lower measurement error than the universal goniome- ter, the standard tool for assessing joint range of motion.
Body Mass Index | The evolution of the variable will be evaluated on days 60 and 120.
  It will be measured by bioelectrical impedance.
Cardiac function | The evolution of the variable will be evaluated on days 60 and 120.
  It will be assessed by monitoring heart rate during exercise, using a chest-strap heart rate monitor.

SECONDARY OUTCOMES:
Upper limb function | The evolution of the variable will be evaluated on days 60 and 120.
  Assessed using the Disabilities of the Arm, Shoulder, and Hand (DASH) questionnaire, in its validated Spanish version.
Wrist and hand pain | The evolution of the variable will be evaluated on days 60 and 120.
  Measured using a Visual Analogue Scale
Sleep quality | The evolution of the variable will be evaluated on days 60 and 120.
  Used as an indicator of quality of life and assessed with the Pittsburgh Sleep Quality Index (PSQI) and accelerometry.
Level of body awareness | The evolution of the variable will be evaluated on days 60 and 120.
  Measured with the Body Awareness Questionnaire
Mindfulness or dispositional mindfulness values | The evolution of the variable will be evaluated on days 60 and 120.
  Measured using the Mindfulness Attention Awareness Scale and used as an indicator of psychological well-being.
Anxiety level | The evolution of the variable will be evaluated on days 60 and 120.
  Measured with the Hamilton Anxiety Scale, an anxiety scale with good psychometric properties that has been used in previous aikido studies.
Positive and negative affect values | The evolution of the variable will be evaluated on days 60 and 120.
  Measured using the Positive Affect Negative Affect Schedule, a test previously used in aikido interventions to assess their effect on the psychological state of practitioners.

CONTACTS AND LOCATIONS:
Locations (1):
- Catholic University of Murcia (UCAM), Murcia, Murcia, Spain

IPD SHARING:
Plan to Share IPD: No